CLINICAL TRIAL: NCT02061111
Title: NeoThyr - the Role of Mitochondria-dysfunction in Newborns of Mothers With Autoimmune Thyroid Disease
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Collaborators: University of Southern Denmark (Other); Region Zealand (Other)
Responsible Party: Principal Investigator, Julie K. G. Stryhn, MD, Naestved Hospital
Other Study IDs: SJ-361
Record Dates: First submitted 2014-01-22; First posted 2014-02-12 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Subclinical Hypothyroidism; Autoimmune Thyroid Disease; Alteration of Mitochondrial Membrane
Keywords: Mitochondria Function; TPO-antibodies; Subclinical Thyroid Disease; Thyroid Disease In Pregnancy; Children´s Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from 77 women and their children´s cords will be stored for 15 years for supplementary analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subclinical thyroid disease: 26 pregnant women with subclinical hypothyroidism and/orTPO-antibodies, and their offspring.
- Healthy controls: 51 pregnant women without thyroid disease or any other metabolic disorders, and their offspring.

SUMMARY:
Previously, studies have shown that children of women with thyroid autoantibodies experience more birth complications and poorer health in their first days. Studies have also shown later signs of cognitive developmental challenges (risk of attention deficit/hyperactivity problems) among children of mothers with autoimmune thyroid disease and/or subclinical hypothyroidism. In Denmark there is no formalized screening or treatment of subclinical thyroid disease - with or without Thyroid Peroxidase Antibodies (TPO-antibodies) - among pregnant women.

The hypothesis of this study is that the offspring of women with subclinical thyroid disease have a mitochondria-dysfunction which leads to more complications during birth, poorer health and well-being in the early childhood. The investigators will test this by recruiting mothers by a blood sample in the third trimester of pregnancy, screen the cord blood at birth and later on test the children with Bayley test two times in the early childhood.

DETAILED DESCRIPTION:
Prior to a planned caesarean section, maternal blood samples are drawn and at the cesarean, cord blood samples are drawn, when the cord is clamped and cut. Thyrotropin, free T3, free T4, anti-TPO and lipids are measured on maternal as well as cord samples. Flow cytometry is performed to measure mitochondrial function. At age 6 months and 15 months the child´s development is evaluated by the Bayley-III test.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy, clinically healthy

Exclusion Criteria:

* Twin-pregnancy, metabolic disorder, medication or other diseases with a potential adverse impact on the pregnancy and fetus

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be selected among pregnant women in region Zealand that will give birth by cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Mitochondrial function | Delivery
  Maternal and cord blood. Analyses will be run by flow cytometry and qPCR

SECONDARY OUTCOMES:
Perinatal complications | At birth
  Number of children in each group with abnormal apgar score, cord pH, need of CPAP, resuscitation, low blood sugar, cramps, death
Well-being | Age 0-15 months
  Number of children in each group that have been admitted to the hospital due to icterus or metabolic disease
Weight (kg) | Age 0-15 months
  Differences between the two groups
Length (cm) | Age 0-15 months
  Differences between the two groups
Head circumference (cm) | Age 0-15 months
  Differences between the two groups
Motor development | Age 6 and15 months
  Differences between the two groups, evaluated by Bayley test
Cognitive development | Age 6 and 15 months
  Differences between the two groups, evaluated by Bayley test
Language | Age 6 and 15 months
  Differences between the two groups, evaluated by Bayley test
Birth complications | Birth
  Number of birth complications in the two groups in terms of postpartum hemorrhage >=500 ml
Social/emotional behavior | Age 12 months
  Differences between the two groups, evaluated by ASQ:SE

CONTACTS AND LOCATIONS:
Overall Officials: Julie Stryhn, MD, Principal Investigator — Naestved Hospital; Peter Gæde, MD, Study Chair — Slagelse Hospital
Locations (1):
- Gynaecologic-Obstetrics Department Naestved Hospital, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No